CLINICAL TRIAL: NCT05178472
Title: Part A: Effect of Prophylactic Vertebroplasty Combined With Radiation Therapy for Spine Metastatic Cancer Patients With Indeterminate Lesion (SINS Criteria)
Brief Title: Vertebroplasty With Radiation Therapy for Spine Metastatic Cancer Patients With Indeterminate Lesion (SINS Criteria)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dukagjin Blakaj, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20048; NCI-2020-13764 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Spine
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Immunotherapy; Adjuvants, Immunologic; Radiosurgery; Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (vertebroplasty) (Experimental): Patients undergo vertebroplasty and, 2-4 weeks later, undergo SRS over 1-3 fractions depending upon the number of affected vertebral bodies. Patients also receive standard of care immunotherapy IV every 2 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Immunotherapy; Radiation: Stereotactic Radiosurgery; Procedure: Vertebroplasty
- Arm II (no vertebroplasty) (Active Comparator): Patients receive standard of care immunotherapy IV every 2 weeks for up to 6 months and undergo SRS over 1-3 fractions depending upon the number of affected vertebral bodies in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Immunotherapy; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Immunotherapy — Receive SOC immunotherapy
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy
Procedure: Vertebroplasty — Undergo vertebroplasty
  Arms: Arm I (vertebroplasty)

SUMMARY:
This clinical trial studies the side effects of stereotactic radiosurgery and how well it works with or without vertebroplasty, separation surgery, or immunotherapy in patients with cancer that is radiation resistant and has spread to the spine (spinal metastases). Spinal metastases are rapidly progressive, have poor prognosis, are extremely difficult to treat, and can effect patient quality of life and overall health. Immunotherapy is a type of standard of care therapy to boost or restore the ability of the immune system to fight cancer. Stereotactic radiosurgery is a type of external radiation therapy that uses special equipment to position the patient and precisely give a single large dose of radiation to a tumor. A vertebroplasty is a procedure used to repair a bone in the spine that has a break caused by cancer, osteoporosis, or trauma. The purpose of this trial is to test different combinations of immunotherapy, stereotactic radiosurgery, and surgery to improve overall survival and quality of life in patients with spinal metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall efficacy and safety of stereotactic radiosurgery (SRS) with or without vertebroplasty or separation surgery in patients with radiation resistant histologies metastatic to the spine with or without concurrent immunotherapy with PD1 blockade.

SECONDARY OBJECTIVES:

I. To assess 6 month vertebral compression fracture (VCF) rate. II. To assess local control (LC) and distant disease control rates. III. To assess the progression free survival (PFS). IV. To assess the overall survival (OS). V. To assess potential vertebral compression fracture (VCF) risk in cancer patients with spinal metastases (SM).

VI. To assess changes in pain from baseline with patient reported measures, medication changes, and quality of life (QoL) measures.

EXPLORATORY OBJECTIVES:

I. To assess changes in immune-stimulatory effect via Trex1 relative to radiation dose.

II. To evaluate whether changes in Trex1 correlates with PD-L1 expression. III. To validate known molecular signatures predicting metastatic potential and molecular mechanisms that have previously been documented.

IV. To develop novel molecular biomarker signatures that predict local spinal metastasis control.

V. To evaluate molecular signatures at the time of spinal metastasis, and potentially define the "molecular evolution" of a tumor after treatment.

OUTLINE:

INDETERMINATE COHORT: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo vertebroplasty 2-4 weeks later, undergo SRS over 1-3 fractions depending upon the number of affected vertebral bodies in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo SRS over 1-3 fractions depending upon the number of affected vertebral bodies in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and older with indeterminate Spine Metastasis.
* All patients with metastatic radiation resistant histologies to the spine (such as Non-small cell Lung cancer, Melanoma, Colorectal, Sarcoma, head and neck, Esophageal, Gallbladder, Liver, Pancreatic, Prostate, Breast, Thyroid, Renal Cell Carcinoma)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Disease visualized by CT or MRI
* Prior radiation therapy will be allowed at the discretion of the Radiation Oncologist based on current standard operating procedures.
* Tumor tissue from the core biopsy or resected site of disease will be collected, if available for biomarker analyses.
* Four or less consecutive spinal segments involved by tumor. Or four or less separate spinal tumor targets with a minimum of one vertebral body separation
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaire in either English or Spanish. The baseline assessment must be completed within required timelines. Inability (illiteracy in English or Spanish, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible

Exclusion Criteria:

* Patients < 18 years of age
* Inability to get a standard MRI or CT myelogram for radiation treatment target delineation
* Patients with prior radiation to the spinal segment to be treated may be included if the radiation dose can be delivered safely, per the treating radiation oncologist.
* Patients with symptomatic spinal cord compression requiring emergent surgery
* Pregnant or lactating women
* Systemic therapy or immunosuppressive medications, excluding immunotherapy, within 3-14 days of radiation treatment, at the discretion of the treating radiation oncologist .
* Patients with stable or unstable lesions based on SINS criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vertebral compression fracture (VCF) rate | At 6 months
  Will be summarized for all patients overall and by each cohort. The confidence interval of the overall VCF rate within 6 months will be calculated using binomial exact test for each cohort.
Local control | At 6 months
  Will be summarized for all patients overall and by each cohort. Will be summarized using Kaplan-Meier survival analysis.

SECONDARY OUTCOMES:
Overall survival | Up to 1 year
  Will be summarized for all patients overall and by each cohort. Will be summarized using Kaplan-Meier survival analysis.
Progression-free survival | Up to 1 year
  Will be summarized for all patients overall and by each cohort. Will be summarized using Kaplan-Meier survival analysis.
Objective response rate | Up to 1 year
  Will be summarized for all patients overall and by each cohort.
Change in health-related quality of life | Baseline up to 1 year
  Will be summarized for all patients overall and by each cohort and estimated using the linear mixed model for repeated measures for each group and overall.
Abscopal effects | Up to 1 year
  Will be summarized for all patients overall and by each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Dukagjin M Blakaj, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu